CLINICAL TRIAL: NCT03988335
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2a Study to Evaluate the Efficacy and Safety of RIST4721 in Subjects With Palmoplantar Pustulosis
Brief Title: A Study to Evaluate RIST4721 in Palmoplantar Pustulosis (PPP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aristea Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RIST4721-201
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Palmoplantar Pustulosis
Keywords: PPP
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIST4721 (Experimental): RIST4721 as once-daily 300mg oral solution for 28 days.
  Interventions: Drug: RIST4721
- Placebo (Placebo Comparator): Placebo as once-daily 300mg oral solution for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RIST4721 — RIST4721 oral solution
  Arms: RIST4721
Drug: Placebo — Placebo oral solution
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Phase 2a Study to Evaluate the Efficacy and Safety of RIST4721 in Subjects with Palmoplantar Pustulosis

ELIGIBILITY:
Inclusion Criteria:

* At least a 6-month history of PPP as defined by the presence of pustules on palms and/or soles, but without evidence of infection on palms and soles
* Moderate or severe PPP, as defined by Palmoplantar Pustulosis Psoriasis Area and Severity Index (PPPASI) ≥8 and Palmoplantar Pustulosis Physician Global Assessment (PPPGA) ≥3 at Day -1, and a minimum of 8 fresh pustules at screening (fresh pustule count on both right/left palms and soles) and 20 fresh pustules at Day -1 (fresh pustule count on both right/left palms and soles)
* Males and females must be willing to use birth control as indicated

Exclusion Criteria:

* Moderate to severe psoriasis, as defined by plaque psoriasis covering ≥10% of total Body Surface Area (BSA) at Day -1
* Subject is known to have an immune deficiency or is immunocompromised
* Positive test for hepatitis, human immunodeficiency virus (HIV) or tuberculosis
* Use of topical therapies for PPP within 2 weeks of Day -1 and/or systemic therapies for PPP within 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- Canada (12):
  - Kirk Barber Research, Calgary, Alberta
  - Alberta DermaSurgery Centre, Edmonton, Alberta
  - CARe Clinic (Central Alberta Research Clinic), Red Deer, Alberta
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Brunswick Dermatology Center, Fredericton, New Brunswick
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Dr. Lyne Giroux Medicine Professional Corporation, Greater Sudbury, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - York Dermatology Center, Richmond Hill, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Dre Angelique Gagne-Henley MD Inc., Saint-Jérôme, Quebec
- Germany (5):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Rothhaar Studien GmbH, Berlin
  - Hautarztpraxis Dr. Niesmann & Dr. Othlinghaus, Bochum
  - MensingDerma research GmbH, Hamburg
  - Hautarztpraxis Dr. Wilfried Steinborn, Straubing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bissonnette R, Maari C, Tsianakas A, Reid D, McCutchan S, Baumgartner S, Mackay J, Bhakta N. A Randomized, Double-Blind, Placebo-Controlled, Phase 2a Study to Evaluate the Efficacy and Safety of RIST4721 in Subjects with Palmoplantar Pustulosis. Dermatol Ther (Heidelb). 2021 Dec;11(6):2179-2193. doi: 10.1007/s13555-021-00632-7. Epub 2021 Oct 30. PMID 34716902
- See also: A Randomized, Double-Blind, Placebo-Controlled, Phase 2a Study to Evaluate the Efficacy and Safety of RIST4721 in Subjects with Palmoplantar Pustulosis — http://link.springer.com/content/pdf/10.1007/s13555-021-00632-7.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects must have at least a 6-month history of PPP and have moderate or severe PPP.
Groups:
- RIST4721: Subjects were randomized to receive RIST4721 300 mg oral solution once daily for 28 days.
- Placebo: Subjects were randomized to receive Placebo oral solution once daily for 28 days.
Period: Overall Study
Arm/Group | RIST4721 | Placebo
Started | 16 | 19
Completed | 14 | 18
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who were randomized to either RIST4721 or Placebo
Groups:
- RIST4721: This arm was randomized to receive 300 mg of RIST4721 once daily for 28 days.
- Placebo: This arm was randomized to receive placebo once daily for 28 days.
- Total: Total of all reporting groups
Arm/Group | RIST4721 | Placebo | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 19 | 34
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 16 | 17 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 11 | 12 | 23
  Germany | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Log Transformed Ratio of Postbaseline Fresh Pustule Count at Day 28 to Baseline
Description: Relative change from baseline in fresh pustule count at Day 28
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Log transformed ratio
Groups:
- RIST4721 300 mg: RIST4721 300 mg (mITT Analysis Set)
- Placebo: Placebo (mITT Analysis Set)
Arm/Group | RIST4721 300 mg | Placebo
Number analyzed (Participants) | 14 | 18
Log transformed ratio | 0.86 (0.692) | 0.53 (0.561)
Statistical Analysis 1: Comparison: RIST4721 300 mg vs Placebo; Test type: Other — The primary endpoints were first tested at alpha of 10% (2-sided). If the larger p-value was less than 10% (2-sided), both primary endpoints were to be declared statistically significant. If the larger p-value was greater than 10%, but the smaller p-value was less than 5% (2-sided), then the primary endpoint with the smaller p-value was to be declared statistically significant; p = 0.24, Hochberg's method

2. Primary Outcome: Log Transformed Ratio of Postbaseline Total Pustule Count at Day 28 to Baseline
Description: Relative change from baseline in total pustule count at Day 28
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Log transformed ratio
Arm/Group | RIST4721 300 mg | Placebo
Number analyzed (Participants) | 14 | 18
Log transformed ratio | 0.99 (0.667) | 0.96 (0.672)
Statistical Analysis 1: Comparison: RIST4721 300 mg vs Placebo; Test type: Other — The primary endpoints were first tested at alpha of 10% (2-sided). If the larger p-value was less than 10% (2sided), both primary endpoints were to be declared statistically significant. If the larger p-value was greater than 10%, but the smaller p-value was less than 5% (2-sided), then the primary endpoint with the smaller p-value was to be declared statistically significant; p = 0.804, Hochberg's method

ADVERSE EVENTS:
Time Frame: From ICF signature to end of study participation (approximately 73 days)
Groups:
- RIST4721 300 mg: All subjects who received at least one dose of RIST4721 300 mg (Safety Analysis Set).
- Placebo: All subjects who received at least one dose of Placebo (Safety Analysis Set).
Arm/Group | RIST4721 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/19
Other Adverse Events (participants affected / at risk) | 13/15 | 7/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIST4721 300 mg (N=15) | Placebo (N=19)
Fatigue (General disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bacterial test (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 3 (3) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 2 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT03988335/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03988335/SAP_001.pdf